CLINICAL TRIAL: NCT03031262
Title: Efficacy and Safety of Chidamide in CBF Leukemia
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIT2016007（Chidamide）
Record Dates: First submitted 2017-01-12; First posted 2017-01-25 (Estimated); Last update posted 2025-05-30 (Actual); Status verified 2025-02

CONDITIONS: AML
MeSH Terms: interventions — Cytarabine; N-(2-amino-5-fluorobenzyl)-4-(N-(pyridine-3-acrylyl)aminomethyl)benzamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High Dose of Cytarabine (Active Comparator): CBF Patients who reach CR after reduction therapy receive high dose of cytarabine.
  Interventions: Drug: Cytarabine
- HDAC + Chidamide (Experimental): CBF Patients who reach CR after reduction therapy receive high dose of cytarabine plus chidamide.
  Interventions: Drug: Cytarabine; Drug: Chidamide

INTERVENTIONS:
Drug: Cytarabine — Cytarabine at a dose of 3g/㎡/d on the first, third and fifth day.
  Other Names: HDAC
Drug: Chidamide — Chidamide at a dose of 20mg/d twice a week for 3 months.
  Arms: HDAC + Chidamide

SUMMARY:
In this open-label, randomized, prospective clinical trial, CBF acute myeloid leukemia (AML) patients who have reached CR are randomised into two groups and receive high-dose cytarabine (HDAC) or high-dose cytarabine plus chidamide.The safety and efficacy of chidamide is evaluated.

DETAILED DESCRIPTION:
In this open-label, randomized, prospective clinical trial, CBF AML(including AML1-ETO or CBF-MYH11 mutated patients) patients who have reached CR are randomised into two groups and receive HDAC or high dose of cytarabine plus chidamide.

In experimental group, patients receive cytarabine at a dose of 3g/㎡/d on the first, third and fifth day and chidamide at a dose of 20mg/d twice a week for 3 months.Patients in control group only receive cytarabine at the same dose.

The safety and efficacy of chidamide is evaluated. The primary outcome is relapse-free survival rate after treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Age of 14 to 55 years old;
2. Patients that meet the diagnostic criteria(WHO 2008 criteria) of AML (except APL subtypes) and with AML1-ETO or CBF-MYH11 mutation.
3. Reached CR after induction regimen.
4. ECOG score of ≤ 2;
5. Patients with eligible laboratory examination including liver,renal and heart function.
6. Adult patients are willing to participate in the study and sign the informed consent by themselves or by their immediate family. Patients under 18 years old willing to participate should have their legal guardians sign the informed consent.

Exclusion Criteria:

1. Secondary leukemia.
2. Patients had other tumor at active stage or had received radiotherapy or chemotherapy in the last 6 months due to other tumor.
3. Patients with other blood diseases(for example, haemophiliacs) are excluded.However, patients with abnormal blood count, but with undiagnosed MDS or MPD patients are included.
4. Acute panmyelosis with myelofibrosis and myeloid sarcoma patients;
5. With BCR-ABL fusion gene;
6. Pregnant or lactating women;
7. With ineligible renal or liver function;
8. With active cardiovascular disease;
9. Severe infection disease including uncured tuberculosis pulmonary aspergillosis;
10. AIDS;
11. Patients had central nervous system involvement when they were diagnosed as AML.
12. Patients with epilepsy or dementia or other mental disease who couldn't understand or follow the research.
13. Drugs, medical, mental or social situation may distract patients from following the research or being evaluated the results.
14. Patients with other factors which were considered unsuitable to participate in the study by the investigators.

Ages: 14 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 250 (Estimated)
Dates: Start 2017-02-08 (Actual); Primary Completion 2025-04-10 (Actual); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Relapse-Free Survival Rate (RFS) | Within 5 years after randomization
  RFS is defined as the time from the date of complete remission (CR) after entry in this trial until the date of documented relapse or death for CBF positive leukemia patients who achieve CR.

SECONDARY OUTCOMES:
Non-relapse Mortality | through treatment completion, an average of 5 months
Overall Survival Rate (OS) | Within 5 years after randomization
Cumulative incidence of relapse | Within 5 years after randomization

CONTACTS AND LOCATIONS:
Overall Officials: Jianxiang Wang, Dr, Principal Investigator — Institute of Hematology & Blood Diseases Hospital, China
Locations (1):
- Institute of Hematology & Blood Diseases Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No